CLINICAL TRIAL: NCT05387265
Title: A Phase 1/1b, Open-label, Dose-finding, First-in-human Study to Evaluate the Safety and Antitumor Activity of CX-904, an EGFR-targeted T-cell Engager in Advanced Solid Tumors (CTMX-904-101)
Brief Title: A Trial to Find Safe and Active Doses for an Investigational Drug, CX-904, for Patients With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: CytomX Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTMX-904-101
Record Dates: First submitted 2022-05-19; First posted 2022-05-24 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CX-904 (Experimental)
  Interventions: Drug: CX-904

INTERVENTIONS:
Drug: CX-904 — CX-904 is a T-cell engaging bispecific Probody® candidate against Epidermal Growth Factor Receptor (EGFR) and CD3.

SUMMARY:
The purpose of this first-in-human study, CTMX-904-101, is to characterize the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD) and antitumor activity of CX-904 in adult subjects with metastatic or locally advanced unresectable solid tumors.

DETAILED DESCRIPTION:
This is a first-in-human study evaluating the safety, tolerability, and activity of CX-904, a conditionally activated T-cell bispecific to EGFR and CD3. The design includes single patient cohorts and a 3+3 design. Escalating dose increments will be determined in discussion with a Safety Review Committee.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic or locally advanced unresectable solid tumor. Must have received prior standard therapy.
* Measurable disease per RECIST 1.1
* Eastern Cooperative Oncology Group performance status of 0 or 1
* Adequate baseline laboratory values
* Patients of childbearing potential or those with partners of childbearing potential must agree to use a highly effective method of birth control from signing the ICF, and for a period of 30 days after the last dose of CX-904.
* Additional inclusion criteria may apply

Exclusion Criteria:

* History of malignancy that was active within the previous 2 years. Exceptions include localized cancers that are not related to the current cancer being treated, that are considered to have been cured, and in the opinion of the Investigator, present a low risk of recurrence
* Screening electrocardiogram demonstrating a mean QTcF value > 480 msec; a screening echocardiogram with left ventricular ejection fraction (LVEF) < 50%
* Serious concurrent illness
* History of or current active autoimmune diseases
* History of myocarditis regardless of the cause
* Pregnant or breast feeding
* Additional exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2022-05-16 (Actual); Primary Completion 2025-06-04 (Actual); Study Completion 2025-06-04 (Actual)

PRIMARY OUTCOMES:
Patients Experiencing Dose-limiting Toxicity | 12 months
  The number of patients experiencing a dose-limiting toxicity (DLT) as defined in the protocol at any dose level during dose escalation.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 30 months
  ORR is the proportion of patients in the efficacy-evaluable population with a best response of Complete Response (CR) or Partial Response (PR) based on Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 by Investigator assessment.
Duration of Response (DOR) | 30 months
  The time from the first documentation of CR or PR (based on RECIST v1.1) that is subsequently confirmed to the first documentation of disease progression or death due to any cause on study, whichever occurs first.
Investigator-assessed Progression-Free Survival (PFS) | 30 months
  The time from the date of the first dose of study treatment until documentation of objective tumor progression based on RECIST v1.1 or until death due to any cause, whichever occurs first.
Disease Control Rate (DCR) | 30 months
  DCR is defined as the rate of confirmed CR, PR, and stable disease (SD) as per RECIST v1.1.
Overall Survival (OS) | 30 months
  The time from treatment initiation until death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Monika Vainorius, M.D., Study Director — CytomX Therapeutics, Inc
Locations (5):
- United States (5):
  - Sarah Cannon Research Institute at HealthONE, Denver, Colorado
  - Sarah Cannon Research Institute, LLC, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - South Texas Accelerated Research Therapeutics, LLC, San Antonio, Texas
  - Virginia Cancer Specialist, Fairfax, Virginia